CLINICAL TRIAL: NCT03555721
Title: CytID Analysis of Oral Lesions
Status: Terminated | Type: Observational
Why Stopped: low subject recruitment
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Mark Nichols, Clinical Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-GEN-17-1067
Record Dates: First submitted 2018-05-29; First posted 2018-06-13 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Oral Cavity Cancer; Oropharyngeal Cancer
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms | interventions — Diagnosis, Oral; Biopsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Oral examination followed by biopsy, CytID, and hpvID: Identification of oral lesions with oral examination with both incandescent light and fluorescent light (OralID), and subsequent testing of suspicious oral lesions with biopsy, CytID, and hpvID
  Interventions: Other: Oral examination with incandescent light; Other: Oral examination with OralID; Diagnostic Test: Biopsy; Diagnostic Test: CytID; Diagnostic Test: hpvID

INTERVENTIONS:
Other: Oral examination with incandescent light — Suspicious oral lesions will be identified by oral examination with incandescent light.
Other: Oral examination with OralID — OralID uses a proven, optically based fluorescence technology that provides the clinician an aid in visualization of oral cancer, pre-cancer and other abnormal lesions.
Diagnostic Test: Biopsy — Tissue will be collected to identify pre-cancerous or cancerous cells
Diagnostic Test: CytID — CytID™ is an adjunctive process that is a noninvasive, pain-free, chair-side procedure for assessment of suspicious oral cavity lesions using a brush swab. The test is based on an objective measure of gross changes in the nuclear DNA content of oral epithelial cells; thereby, providing information about the pre-cancerous or cancerous state of a lesion.
Diagnostic Test: hpvID — hpvID™ testing can detect all major HPV types and shows the current HPV status of the patient. This provides additional clinical information to correlate and compare hpvID™ trends with routine standard of care biopsy or cytology results.

SUMMARY:
The purpose of this study is to correlate the results from a standard of care biopsy with CytID™ and hpvID™ swab tests for potentially premalignant and malignant oral lesions. The biopsy is considered standard of care and will be performed regardless of the patient's enrollment in the study. The study-related data gathering will not influence the treatment decisions of the clinician.

ELIGIBILITY:
Inclusion Criteria:

* Receive care at the Avenue 360 Health and Wellness Clinic, a not for profit dental clinic in the Montrose area of Houston
* Present with a potentially malignant oral lesion (PMOL) for whom a biopsy is deemed necessary

Exclusion Criteria:

* Do not receive care at the Avenue 360 Health and Wellness Clinic, a not for profit dental clinic in the Montrose area of Houston
* Do not present with a potentially malignant oral lesion (PMOL) for whom a biopsy is deemed necessary

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who receive care at the Avenue 360 Health and Wellness Clinic, a not for profit dental clinic in the Montrose area of Houston (a federally qualified health center).
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Number of participants for whom biopsy and CytID results both indicate presence of malignant or premalignant oral lesions | day 1 (at the time of oral examination)
Number of participants for whom biopsy indicates presence of malignant or premalignant oral lesions and hpvID indicates presence of HPV | day 1 (at the time of oral examination)
Number of participants for whom biopsy results, but not CytID results, indicate presence of malignant or premalignant oral lesions | day 1 (at the time of oral examination)
Number of participants for whom CytID results, but not biopsy results, indicate presence of malignant or premalignant oral lesions | day 1 (at the time of oral examination)
Number of participants for whom biopsy does not indicate presence of malignant or premalignant oral lesions, but hpvID indicates presence of HPV | day 1 (at the time of oral examination)
Number of participants for whom biopsy indicates presence of malignant or premalignant oral lesions, but hpvID does not indicate presence of HPV | day 1 (at the time of oral examination)

CONTACTS AND LOCATIONS:
Overall Officials: Clifton M Nichols, DDS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States